CLINICAL TRIAL: NCT05397795
Title: COMPARING TWO PROTOCOLS FOR FINAL OOCYTE MATURATION IN POOR RESPONDERS UNDERGOING GnRH-ANTAGONIST ICSI CYCLES
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DT193
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Infertility
Keywords: Oocyte Maturation; ICSI; poor responders; Trigger; Dual Trigger
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin; Triptorelin Pamoate

STUDY DESIGN:
Intervention Model Description: Before enrollment in the study, all patients will be subjected to routine medical evaluation to make sure of presence of inclusion criteria and absence of exclusion criteria. Then women will be randomized using computer-based randomization (Random Digit Software).
  All included women will undergo a fixed GnRH antagonist protocol of COH.
  At the day of triggering, number of follicles and the number of oocytes expected to be retrieved will be documented and women will be given the trigger according to the randomization done at the enrollment.
  Two main groups will be created depending on the trigger protocol used:
  Group A: 80 subjects will be triggered by 10000 IU of hCG (Choriomon5000 IU; IBSA) given intramuscularly.
  Group B: 80 subjects will be triggered by 10000 IU of hCG (Choriomon5000 IU; IBSA) intramuscular injection in addition to the GnRH agonist triptorelin 0.2 mg (Decapeptyl 0.1 mg; Ferring) subcutaneously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group(A) (Experimental): subjects will be triggered by 10000 IU of hCG (Choriomon5000 IU; IBSA) given intramuscularly.
  Interventions: Drug: 10000 IU hCG (Choriomon5000 IU; IBSA)
- Group(B) (Experimental): subjects will be triggered by 10000 IU of hCG (Choriomon5000 IU; IBSA) intramuscular injection in addition to the GnRH agonist triptorelin 0.2 mg (Decapeptyl 0.1 mg; Ferring) subcutaneously.
  Interventions: Drug: 10000 IU hCG (Choriomon5000 IU; IBSA); Drug: Triptorelin 0.2 mg (Decapeptyl 0.1 mg; Ferring)

INTERVENTIONS:
Drug: 10000 IU hCG (Choriomon5000 IU; IBSA) — 10000 IU of hCG (Choriomon5000 IU; IBSA) given intramuscularly
  Other Names: CHORIONIC GONADOTROPHIN 5000 U
Drug: Triptorelin 0.2 mg (Decapeptyl 0.1 mg; Ferring) — GnRH agonist triptorelin 0.2 mg (Decapeptyl 0.1 mg; Ferring) subcutaneously.
  Other Names: TRIPTOFEM 0.1 mg
  Arms: Group(B)

SUMMARY:
Poor ovarian responders (POR) include a significant proportion of women referred for IVF treatments (ranging from 9 to 24 %), most of whom are in late reproductive age.

In fact the live birth rate in the entire POR category is poor (about 6 % per cycle). However patients <40 years have a significantly better prognosis compared to older patients, mainly due to better oocyte quality.Attempts to improve IVF cycle outcomes for poor responders included modifying the steps of ovarian stimulation protocols , such as different luteal phase pretreatments, increasing ovarian stimulation doses, as well as addition of various supplements. So far, most of the modifications had limited success, therefore, optimal protocol for poor responders has remained elusive.

Final oocyte maturation trigger is one of the most important key success factors in assisted reproductive technologies (ARTs). Oocyte maturation refers to a release of meiotic arrest that allows oocytes to advance from prophase I to metaphase II of meiosis. Luteinizing Hormone (LH) surge by dismantling the gap junctions between granulosa cells and oocyte inhibits the flow of maturation inhibitory factors into ooplasm and causes drop in concentration of cAMP. Decreased concentration of cyclic AMP (cAMP) in turn increases concentration of Ca and maturation-promoting factor (MPF), which are essential for the resumption of meiosis in oocyte and disruption of oocyte-cumulus complex triggering follicular rupture and ovulation about 36 h the LH surge.

The aim of the study is to compare the oocyte yield , oocyte quality and the ongoing pregnancy rate between dual trigger treatment (combination of gonadotrophin-releasing hormone (GnRH) agonist and human chorionic gonadotrophin) and human chorionic gonadotrophin alone in PORs undergoing in vitro fertilization/intracytoplasmic sperm injection (IVF-ICSI) cycles using a GnRH-antagonist protocol.

DETAILED DESCRIPTION:
Poor ovarian responders (POR) include a significant proportion of women referred for IVF treatments (ranging from 9 to 24 %), most of whom are in late reproductive age.(1,2) According to the "Bologna criteria", patients are classified as POR based on three conditions: if two or more of the following features are present: 1) advanced maternal age (>40 years); 2) a previous poor ovarian response (cycles cancelled or <3 oocytes with a conventional protocol); 3)an abnormal ovarian reserve test (antral follicle count 5-7 follicles or anti-Mullerian hormone 0.5-1.1 ng/ ml). Two of these criteria are required for a POR diagnosis. In addition, two cycles with POR after maximal stimulation are sufficient to classify a patient as a poor responder even in the absence of other criteria mentioned. (3)

In fact the live birth rate in the entire POR category is poor (about 6 % per cycle).(4,5) however patients <40 years have a significantly better prognosis compared to older patients, mainly due to better oocyte quality.(6) Attempts to improve IVF cycle outcomes for poor responders included modifying the steps of ovarian stimulation protocols , such as different luteal phase pretreatments, increasing ovarian stimulation doses, as well as addition of various supplements. So far, most of the modifications had limited success, therefore, optimal protocol for poor responders has remained elusive.(7)

ESHRE in 2019 stated GnRH antagonists and GnRH agonists are equally recommended for predicted low responders. (8)

Final oocyte maturation trigger is one of the most important key success factors in assisted reproductive technologies (ARTs). Oocyte maturation refers to a release of meiotic arrest that allows oocytes to advance from prophase I to metaphase II of meiosis. Luteinizing Hormone (LH) surge by dismantling the gap junctions between granulosa cells and oocyte inhibits the flow of maturation inhibitory factors into ooplasm and causes drop in concentration of cyclic AMP (cAMP) . Decreased concentration of cAMP in turn increases concentration of Ca and maturation-promoting factor (MPF), which are essential for the resumption of meiosis in oocyte and disruption of oocyte-cumulus complex triggering follicular rupture and ovulation about 36 h the LH surge.(9)

Until now, administering 5000 IU to 10,000 IU of hCG 34-36 h prior to oocyte retrieval remained the standard protocol for the induction of final oocyte maturation in IVF cycles worldwide. Traditionally, human chorionic gonadotropin (hCG) has been the trigger of choice for oocyte maturation due to its molecular and biological similarity with LH.(10)

Gonadotropin-releasing hormone (GnRH) agonists were first suggested for final oocyte maturation by Gonen et al. in 1990, as it is able to trigger endogenous release of both FSH and LH.(11) With a shorter mean duration of LH surge of about 34 hours, it is similar to the natural cycle duration of 48 hours,(12) effectively reducing the incidence of Ovarian Hyperstimulation Syndrome (OHSS) in high responders.(13,14) However, some problems surfaced with the substitution of GnRH-agonists as trigger. The risk of empty follicle syndrome was reported to be increased following isolated GnRH-agonist trigger due to a suboptimal LH surge(15) ,in addition, increased early pregnancy loss and decreased rates of ongoing pregnancy were noted by multiple studies.(16,17) As such, the idea of a dual trigger was developed.(18) Indeed, the hCG component of dual trigger could serve as a rescue trigger in case of poor response to GnRH-agonist, which occurs in about 2.71% of a study population.(19) In combining GnRH-agonist and hCG for the final oocyte maturation , we get the benefits of both. HCG administration alone also does not produce Follicle Stimulating Hormone(FSH) activity, while GnRH-agonist releases an endogenous FSH and LH surge, resulting in a more physiologic response.

In addition, another proposed advantage with dual trigger is potential enhancement of endometrial receptivity by the GnRH-a component. Significant elevation of both isoforms of human GnRH messenger Ribonucleic Acid (mRNA) expression have been detected in the secretory phase of the human menstrual cycle,(20-22) indicating the possible role of these hormones in regulation of endometrial receptivity.(20,23) Specifically, in vitro studies with human extra-villous cytotrophoblasts and decidual stroma cells have demonstrated the ability of GnRH to activate urokinase type plasminogen activator, a key component in decidualization and trophoblast invasion.(24,25) Therefore, inclusion of GnRH-a as part of luteal support regimen has been explored as a mean to improve the implantation rate.

Since its development, multiple investigations have shown the benefits of using a dual trigger for final oocyte maturation in normal responders,(16,26) including an improvement in total number of retrieved oocytes, MII oocytes, rates of embryo implantation, clinical pregnancy, and live birth rates.(27) Evidence from available meta-analysis in 2018 involving four studies including 527 patients found a significantly improved clinical pregnancy rate following dual trigger.(28) However, for poor ovarian responders (PORs), the situation is less clear cut.

ESHRE in 2019 stated that dual triggering is not recommended in normal ovarian responders. However, there was no clear recommendation regarding PORs, giving rise to the need to perform a well-designed randomized controlled trial for the evaluation of dual triggering in PORs. .(29,30)

ELIGIBILITY:
Inclusion Criteria:

1. Women with a spontaneous normal menstrual cycle and a normal uterine cavity.
2. Body mass index (BMI) < 35.
3. Age less than 45.
4. Anti-Mullerian Hormone (AMH) ≤ 1.1 ng/ ml
5. Antral Follicle Count (AFC) ≤ 7 follicles

Exclusion Criteria:

1. Comorbidities including, hypertension, Diabetes Mellitus or other endocrinopathies.
2. Surgically retrieved sperms.
3. Communicating hydrosalpinx.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female In Reproductive Age group
Enrollment: 160 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of metaphase II oocytes retrieved. | On 1 day of oocyte retrieval
  Number of metaphase II oocytes retrieved

SECONDARY OUTCOMES:
Total number of oocytes | On 1 day of oocyte retrieval
  Total number of oocytes
Ratio between number of follicles seen on day of trigger and number of oocytes retrieved | On 1 day of oocyte retrieval
  Ratio between number of follicles seen on day of trigger and number of oocytes retrieved
Maturity index | On 1 day of oocyte retrieval
  Number of metaphase II oocytes retrieved per total number of oocytes retrieved
Fertilization rate | On 1 day after oocyte retrieval
  Number of fertilized oocyte per total number of oocytes retrieved
Cancellation rate | Folliculometry on day 8 revealed no growing follicles, serum estradiol level less than 150 pg/mL on the day of hCG administration, no oocytes were retrieved, or if fertilization failed
  Folliculometry on day 8 revealed no growing follicles, serum estradiol level less than 150 pg/mL on the day of hCG administration, no oocytes were retrieved, or if fertilization failed
Number of obtained embryos | On 1 day after oocyte retrieval
  Number of obtained embryos
Number of transferred embryos | On 1 day of embryo transfer
  Number of transferred embryos
Quality of embryos transferred | On 1 day of embryo transfer
  Quality of embryos transferred using an embryo grading system
Day of transfer | Two to five days after oocyte retrieval
  Day of transfer
Implantation rate | Between the 5th to 6th weeks of gestation.
  Total number of observed gestational sacs divided by the total number of transferred embryos
Chemical pregnancy rate | Fourteen days after embryo transfer
  Transient positive serum beta-hCG level without subsequent development of visible gestational sac.
Clinical pregnancy rates | Between the 5th to 6th weeks of gestation.
  Visualization of the fetal heart beat by ultrasound between the 5th to 6th weeks of gestation.
Ongoing pregnancy rates | 20 weeks of gestation.
  Number of fetuses with heart activity beyond 20 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Mervat Sh EL-Arab, MDPhD, Principal Investigator — mervatsheikhelarab@gmail.com

IPD SHARING:
Plan to Share IPD: Yes
By the end of the study, we will share the data in a supplementary file.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Just after completion of the study and the data will be open accessed
Access Criteria: web address and journals

REFERENCES:
- [Background] Ding N, Liu X, Jian Q, Liang Z, Wang F. Dual trigger of final oocyte maturation with a combination of GnRH agonist and hCG versus a hCG alone trigger in GnRH antagonist cycle for in vitro fertilization: A Systematic Review and Meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2017 Nov;218:92-98. doi: 10.1016/j.ejogrb.2017.09.004. Epub 2017 Sep 14. PMID 28957685